CLINICAL TRIAL: NCT01706289
Title: The Relationship Between Vascular Adhesion Protein-1 and Diabetic Cardiovascular Autonomic Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NTUH20090323HRV
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-09

CONDITIONS: Neuropathy; Peripheral, Autonomic, in Diabetes Mellitus (Manifestation)
Keywords: diabetes; cardiovascular autonomic neuropathy; VAP 1
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diabetic mellitus screen

SUMMARY:
Exploring the relationship between serum VAP-1 and cardiovascular autonomic neuropathy in subjects with type 2 diabetes mellitus

DETAILED DESCRIPTION:
The prevalence of diabetes mellitus is increasing recently, especially in the urban area of developing countries. Subjects with diabetes have higher rate of hospitalization and have higher mortality. Diabetes results in various complications including diabetic retinopathy, nephropathy, neuropathy, and cardiovascular complications. Among these, cardiovascular autonomic neuropathy is one of clinical important complication of diabetes. Diabetic subjects with reduced cardiovascular autonomic function have been shown to strongly associate with an increased risk of silent myocardial ischemia and increased mortality. They also have higher risk of sudden death, intraoperative and perioperative cardiovascular instability. Formation of advanced glycation end product (AGE) and oxidative stress are important causes of diabetic neuropathy. Vascular adhesion protein-1 (VAP-1), an adhesion molecule with an activity of semicarbazide-sensitive amine oxidases (SSAO), which can catalyze endogenous amines to produces corresponding aldehydes, H2O2, and ammonia. We have demonstrated that serum VAP-1 is a source of systemic AGE and oxidative stress, and is associated with nephropathy and atherosclerosis. There are reports demonstrating that subjects with diabetic retinopathy or stroke have higher serum VAP-1. To our best knowledge, there is no report regarding the relationship between serum VAP-1 and neuropathy. In present study, we will measure serum VAP-1 and check cardiovascular autonomic function. We will also explore the relationship between serum VAP-1 and cardiovascular autonomic neuropathy in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus

Exclusion Criteria:

* arrythmia

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: type 2 diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yaun Li, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Douliu, Taiwan